CLINICAL TRIAL: NCT01325376
Title: SKTA iWell21 Clinical Trial Protocol. This is a Randomized Control Trial of 500 Adult Participants Randomized to Two Arms: Control Arm: Self Directed Program (SDP), Intervention Arm: Dynamic On-line Interactive Technology (DOIT)
Brief Title: PH iWell Study to Compare an Online Interactive Technology to Self-directed Care in Overweight or Obese Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SK Telecom Americas, Inc. (Industry)
Collaborators: PeaceHealth Laboratories (Unknown)
Responsible Party: Brigitte Piniewski, MD/Chief Medical Officer, PeaceHealth Laboratories
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SKTA iWell 21
Record Dates: First submitted 2010-10-22; First posted 2011-03-29 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self directed (No Intervention)
  Interventions: Behavioral: Self directed
- Technology assisted health behavior (Active Comparator): The intervention arm will have access to a dynamic online environment with social networking and device data uploads that include activity data, weight data and laboratory data at frequent intervals to nudge optimal health behavior.
  Interventions: Behavioral: Technology assisted health behavior

INTERVENTIONS:
Behavioral: Technology assisted health behavior — Web-based interactive program using an hpod sensor that tracks physical activity as well as biometric parameters into the iWell server and is transmitted to the internet site via the users PC. Also serves as a social networking site.
  Other Names: DOIT Dynamic online interactive technology
  Arms: Technology assisted health behavior
Behavioral: Self directed — Receives support and encouragement with minimal contact. Receives printed lifestyle guidelines with diet and physical activity recommendations.
  Other Names: Standard care
  Arms: Self directed

SUMMARY:
This is a six month lifestyle management study to compare the effects of iWell; a dynamic online interactive technology to a self-directed program in overweight or obese individuals.

The primary aim is to test the hypothesis that dynamic online interactive technology intervention is more effective than self-directed program in obtaining and maintaining weight loss and other biometric improvements.

DETAILED DESCRIPTION:
Optimal health behavior is difficult to sustain over extended periods. This study seeks to demonstrate that technology can be a low cost scaleable solution that will provide the user with sufficient customization and personalization through social networking approaches such that sustainability of optimal health behavior is realized.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years old
* overweight or obese men and women with BMI between 24 and 38, inclusive
* concerned about weight/health (and motivated in losing weight)
* stable medications for past 3 months
* willing/able to use Web-based services
* willingness not to use weight loss medications for the duration of the trial
* able and willing to give informed consent and participate in the interventions
* willing to come to three sessions and visits
* willingness to be randomized to intervention or control group

Exclusion Criteria:

* contraindication to weight loss (e.g., malignancy or other serious illness)
* Type 1 DM and Type 2 DM with other end organ compromise (renal, retinal or other)
* Recent (within 6 months) cardiovascular event (MI or stroke)
* current symptoms of angina
* heart, renal, or liver disease (excluding kidney stone)
* cancer or active neoplasm (excluding skin cancers)
* hyperthyroidism
* mental conditions that would preclude full participation
* prior weight-loss (bariatric) surgery or plan for these procedures
* liposuction surgery in past 12 months or plan for these procedures
* recent weight loss in the past 3 months (>20 lbs)
* use of prescription weight loss medication in 3 months prior to screening
* current use of medications for treatment of psychosis or manic-depressive illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Weight loss from baseline | at 6 months

SECONDARY OUTCOMES:
Blood pressure change from baseline | at 3 months
  Systolic blood pressure and diastolic blood pressure
Triglyceride level change from baseline | at 3 months
  Participants will have a venous draw to determine Triglyceride levels
High density lipoprotein level change from baseline | at 3 months
  Venous draw to determine high density lipoprotein levels
Physical activity adjustment from baseline | at 3 months
  Standardized activity questionaire and activity monitoring device will be used to determine adjustments in activity for each arm
Blood pressure change from baseline | at 6 months
Triglyceride level change from baseline | at 6 months
High density lipoprotein level change from baseline | at 6 months
Physical activity adjustment from baseline | at 6months
  Standardized activity questionaire and activity monitoring device will be used to determine adjustments in activity for each arm

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Piniewski, MD, Principal Investigator — PeaceHealth Laboratories; David Kil, Principal Investigator — SKTelecom Americas
Locations (1):
- PeaceHealth Laboratories, Springfield, Oregon, United States